CLINICAL TRIAL: NCT05181397
Title: A Prospective, Randomized Controlled Study to Compare Efficacy and Safety of Intravenous 8mg/kg Tocilizumab Versus Regular Treatment for Severe Rapid Progressive Interstitial Lung Diseases (RP-ILD) Secondary to Systemic Diseases
Brief Title: The Efficacy and Safety of Tocilizumab for Severe RP-ILD Secondary to Systemic Diseases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JS-2679
Record Dates: First submitted 2021-12-19; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-03

CONDITIONS: Rapid Progressive Interstitial Lung Diseases
MeSH Terms: interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: Participants are planned to be separated into two groups. 68 participants with severe RP-ILD secondary to systemic diseases will be randomly assigned to receive intravenous 8mg/kg tocilizumab or regular treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab (Experimental): Participants in tocilizumab group will receive intravenous 8mg/kg tocilizumab. No Intervention: control, participants in control group will receive regular treatment.
  Interventions: Drug: Tocilizumab
- Control (No Intervention): Participants in control group will receive regular treatment.

INTERVENTIONS:
Drug: Tocilizumab — Participants in tocilizumab group will receive intravenous 8mg/kg tocilizumab.
  Arms: Tocilizumab

SUMMARY:
There is no confirmed drug therapy for RP-ILD. Prognosis is poor of regular treatment. The study is designed to compare efficacy and safety of tocilizumab versus regular treatment in participants with severe RP-ILD secondary to systemic diseases.

DETAILED DESCRIPTION:
RP-ILD, also known as the acute exacerbation of interstitial lung disease, was defined as an acute, clinically significant respiratory deterioration characterized by evidence of new widespread alveolar abnormality on chest imaging or histopathology. It is rapidly progressive and life-threatening. Despite aggressive regular treatments with high-dose glucocorticoids in combination with immunosuppressant drugs such as cyclosporine, tacrolimus, or cyclophosphamide, the post-exacerbation mortality rates remain high. There is no confirmed drug therapy for RP-ILD. Recently, the exacerbation of interstitial lung diseases secondary to systemic diseases was proved to involve many inflammatory responses, so patients are more likely to benefit from immune regulation therapy. Tocilizumab is a monoclonal antibody that inhibits the binding of interleukin-6 (IL-6), a multifunctional cytokine that regulates the immune response and inflammation, to its receptor (IL-6R). The study is designed to compare efficacy and safety of tocilizumab versus regular treatment in participants with severe RP-ILD secondary to systemic diseases.

ELIGIBILITY:
Inclusion Criteria:

RP-ILD, previous or concurrent diagnosis of systemic diseases

Exclusion Criteria:

pregnancy; uncontrolled pulmonary infections; severe cardiovascular, hepatic and renal dysfunction; unstable angina or myocardial infarction; thrombocytopenia； neutrophil reduction； malignant tumor; allergy to tocilizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
The differences of oxygenation index changes between the two groups on day 7, 14, 28 and month 3 after the first dose* | 3 months
  first dose: The tocilizumab group: the tocilizumab administered for the first time; The control group: the maximum dose of glucocorticoid administered for the first time

SECONDARY OUTCOMES:
Time to clinical stability | 3 months
  clinical stability was defined as on the first day that all of the following criteria are simultaneously achieved: (1) Participants can tolerate walking with or without oxygen therapy; (2) no wheeze; and (3) oxygen saturation >88% on room air.
Survival rate after 3 months | 3 months
Length of stay in hospital | 3 months
Length of stay in ICU | 3 months
Changes of dyspnea index | 3 months
The occurrence of adverse events within 1, 3, 7, 14, 28 days and 3 months after the first dose | 3 months
  adverse events: sepsis, treatment-related hyperglycemia, gastrointestinal bleeding, hospital infection
Changes of erythrocyte sedimentation rate, c-reactive protein or ferritin at baseline and on day 3, 7, 14, 28, month 3 after the first dose | 3 months
Computed tomography score | 3 months
Hospitalization cost | 3 months
Re-admission rate | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Xinlun Tian, M.D., Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
The protocol and clinical study report will be shared.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be shared between time of completion of the study and time of publication of the study.
Access Criteria: contact study director Xinlun Tian, M.D. via xinlun_t@sina.com